CLINICAL TRIAL: NCT05019170
Title: Smartphone-based Financial Incentives to Promote Smoking Cessation Among Alaska Native Pregnant Women
Brief Title: Remote Incentives for Smoking Cessation Among AN Pregnant Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not recruit enough patients
Sponsor: University of Vermont (Other)
Collaborators: Alaska Native Tribal Health Consortium (Other); Mayo Clinic (Other)
Responsible Party: Principal Investigator, Diann Gaalema, Associate Professor of Psychiatry, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1558083
Record Dates: First submitted 2021-08-09; First posted 2021-08-24 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Smoking; Smoking Cessation
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Practice Guidelines as Topic

STUDY DESIGN:
Intervention Model Description: The investigators are proposing a two-condition, parallel groups, randomized controlled pilot study of a smartphone-based financial incentives intervention for AN pregnant smokers. The experimental group will receive financial incentives (money loaded onto a debit card) contingent on the remote submission of breath carbon monoxide and saliva cotinine tests indicating smoking abstinence in addition to best practices for promoting smoking cessation (Best Practices + Incentives). The control group will receive best practices alone (Best Practices). The use of a best practices group reflects a real-world comparison condition in that all women will receive the treatment that practitioners in the community are instructed to provide (the 5As + quitline referral) thereby enhancing the ecological validity of the study. Additionally, the investigators will minimize between-subject variability in the participant's exposure to these practices by implementing these treatment components themselves.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best Practices + Incentives group (Experimental): Participants assigned to this condition will receive the best practices treatment plus the financial incentives intervention.
  Interventions: Behavioral: Smartphone-based Financial Incentives; Behavioral: Best Practices
- Best Practices (Active Comparator): Participants assigned to this condition will receive the best practices treatment alone.
  Interventions: Behavioral: Best Practices

INTERVENTIONS:
Behavioral: Smartphone-based Financial Incentives — Financial Incentives - Beginning on the quit date and extending for one week, participants will be required to submit twice daily CO samples. All samples < 6 ppm will be considered negative and those > 6 ppm will be considered positive. Participants will earn incentives for breath tests indicating smoking abstinence, and incentive values will increase with each consecutive negative sample. Following the initial quit week, the schedule of monitoring will be reduced, and incentives will be contingent on submitting a negative saliva cotinine test.
  Other Names: Contingency Management
  Arms: Best Practices + Incentives group
Behavioral: Best Practices — Best Practices- The 2008 Clinical Practice Guidelines for smoking cessation recommends that pregnant smokers be provided with the 5As. Research staff will implement the 5As at assessments that take place during pregnancy.

SUMMARY:
Cigarette smoking during pregnancy increases risk for catastrophic pregnancy complications, growth retardation, other adverse infant health problems, and later-in-life chronic conditions. One group that is particularly at risk for these complications are Alaska Native (AN) women. Prevalence of smoking during pregnancy is disproportionally high among AN women compared to US pregnant women overall (i.e., ~36% and ~13%, respectively) and few smoking-cessation interventions have been evaluated among this population. A substantive barrier to offering evidence-based interventions to AN women is the geographic remoteness of Alaska. The most effective intervention for promoting smoking cessation during pregnancy is financial incentives in which participants earn incentives (e.g., cash) contingent on objective evidence of smoking abstinence. This intervention has been adapted to be delivered entirely through a smartphone meaning that the geographic remoteness of Alaska will not be a barrier with this intervention. Participants submit videos of themselves completing breath and saliva tests, and incentives are then delivered through the application if the tests indicate smoking abstinence. Through a collaboration between the University of Vermont and the Alaska Native Tribal Health Consortium, the goal of this study is to examine the preliminary feasibility and efficacy of this smartphone-based incentives intervention among AN women. Pregnant AN women will be recruited through ads posted on social media. Eligible participants who complete the informed consent process will be randomized to either: Best Practices or Best Practices + Incentives. In the Best Practices condition, participants will receive three brief educational sessions and a referral to the Alaska state quitline. In the Best Practices + Incentives condition, participants will receive the same education sessions and quitline referral, plus financial incentives contingent on the smartphone-based testing of breath and saliva specimens indicating abstinence from recent smoking. Outcomes will include point prevalence smoking abstinence at assessments conducted in late pregnancy and 4-, 8-, 12-, and 24-weeks postpartum, continuous abstinence during antepartum and postpartum, and perceived barriers and facilitators of treatment engagement. Overall, this project has the potential to address disparities in access to efficacious, evidence-based smoking cessation treatments among AN pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* report being smokers at the time they learned of the current pregnancy
* report smoking in the 7 days prior to completing their preliminary eligibility screening
* < 25 weeks pregnant
* speak English
* own a smartphone (Android or iOS)
* self-report as an Alaska Native
* current smoker as verified by saliva cotinine test

Exclusion Criteria:

* current or prior mental or medical condition that may interfere with study participation
* smoke marijuana more than once each week and not willing to quit (marijuana smoking can inflate breath CO)
* exposed to unavoidable occupational sources of CO (e.g., car mechanic)
* report currently receiving opioid maintenance therapy (e.g., methadone, buprenorphine)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Late Pregnancy Quit Rate | 28 weeks gestation through date of delivery
  Point prevalence smoking abstinence (defined as a cotinine-negative saliva test AND self-reported no smoking in the past seven days)

SECONDARY OUTCOMES:
Early Pregnancy Quit Rate | One month after participant's enrollment date
  Point prevalence smoking abstinence (defined as a cotinine negative saliva test AND self-reported no smoking in the past seven days)
4-Week Postpartum Quit Rate | 4 weeks following the date that participants deliver their infant
  Point prevalence smoking abstinence (defined as a cotinine-negative saliva test AND self-reported no smoking in the past seven days)
8-Week Postpartum Quit Rate | 8 weeks following the date that participants deliver their infant
  Point prevalence smoking abstinence (defined as a cotinine-negative saliva test AND self-reported no smoking in the past seven days)
12-Week Postpartum Quit Rate | 12 weeks following the date that participants deliver their infant
  Point prevalence smoking abstinence (defined as a cotinine-negative saliva test AND self-reported no smoking in the past seven days)
24-Week Postpartum Quit Rate | 24 weeks following the date that participants deliver their infant
  Point prevalence smoking abstinence (defined as a cotinine-negative saliva test AND self-reported no smoking in the past seven days)
Longest Duration of Abstinence (LDA) | LDA will be measured from participant's date of enrollment in the study to 24-weeks postpartum
  Consecutive days of no smoking using biochemical verification (cotinine-negative saliva at the formal assessments) plus self-report (cigarettes per day from enrollment to 24 weeks postpartum reported during timeline follow-back conducted over the phone)

CONTACTS AND LOCATIONS:
Overall Officials: Diann Gaalema, PhD, Principal Investigator — University of Vermont
Locations (2):
- United States (2):
  - Alaska Native Tribal Health Consortium, Anchorage, Alaska
  - University of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurti AN, Tang K, Bolivar HA, Evemy C, Medina N, Skelly J, Nighbor T, Higgins ST. Smartphone-based financial incentives to promote smoking cessation during pregnancy: A pilot study. Prev Med. 2020 Nov;140:106201. doi: 10.1016/j.ypmed.2020.106201. Epub 2020 Jul 9. PMID 32652133

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/70/NCT05019170/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/70/NCT05019170/ICF_001.pdf